CLINICAL TRIAL: NCT03792256
Title: A Phase 1 Study of Palbociclib (IND#141416), A CDK 4/6 Inhibitor, in Combination With Chemotherapy in Children With Relapsed Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LL)
Brief Title: Palbociclib in Combination With Chemotherapy in Treating Children With Relapsed Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AINV18P1; NCI-2019-02774 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-11-29; First posted 2019-01-03 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Lymphocytic; Lymphoblastic Lymphoma; T-cell Lymphoma; T-cell Leukemia; Recurrent Disease; Acute Leukemia
MeSH Terms: conditions — Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell; Leukemia, T-Cell; Recurrence | interventions — palbociclib; Cytarabine; Methotrexate; Hydrocortisone; Doxorubicin; Prednisolone; Vincristine; pegaspargase; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Palbociclib) (Experimental): Patients receive Palbociclib 50 mg/m^2 (starting dose with maximum dose of 100 mg) PO (or via NG-tube) once daily on Days 1-21; Intrathecal cytarabine (IT ARAC) age-based dosing on Day 1, Doxorubicin 60 mg/m^2 IV push or infusion over 1-15 min on Day 4; Prednisone or prednisolone 40 mg/m^2 PO divided BID or TID on days 4-31; Vincristine 1.5 mg/m^2 (maximum dose 2 mg) IV push or mini-bag per institutional policy on days 4, 11, 18, and 25; and Pegaspargase 2500 IU/m^2 IV over 1-2 hours on Days 5, and 18. If CNS3 leukemia is present, patients receive Intrathecal Triple Therapy (ITT) age-based dosing on days 4, 11, 18, and 25. Patients known to be CNS3 at study entry may receive ITT on Day 1 rather than IT ARAC. If CNS1 and 2 leukemia present, patient receive Methotrexate (IT MTX) age-based dosing on Days 18 and 32. Treatment will be given for one cycle, 32 days, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palbociclib; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Doxorubicin; Drug: Prednisolone; Drug: Vincristine; Drug: Pegaspargase; Drug: Prednisone

INTERVENTIONS:
Drug: Palbociclib — Given PO (or via NG- tube)
Drug: Cytarabine — Given intrathecally (IT)
Drug: Methotrexate — Given intrathecally (IT)
Drug: Hydrocortisone — Given IT
Drug: Doxorubicin — Given intravenously (IV)
Drug: Prednisolone — Either prednisone or prednisolone is given PO
Drug: Vincristine — Given IV
Drug: Pegaspargase — Given IV
Drug: Hydrocortisone — Given intrathecally (IT)
Drug: Prednisone — Either prednisone or prednisolone is given PO

SUMMARY:
AINV18P1 is a Phase 1 study where palbociclib will be administrated in combination with a standard re-induction platform in pediatric relapsed Acute Lymphoblastic Leukemia (ALL) and lymphoblastic lymphoma (LL). LL patients are included because the patient population is rare and these patients are most commonly treated with ALL regimens. The proposed palbociclib starting dose for this study will be 50 mg/m^2/day for 21 days.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of palbociclib administered in combination with re-induction chemotherapy in pediatric patients with relapsed B- or T-lineage ALL/LL.

II. To define and describe the toxicities of palbociclib administered on this schedule.

III. To characterize the pharmacokinetics of palbociclib in pediatric patients with relapsed B- or T-lineage ALL/LL.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of palbociclib in combination with chemotherapy for children with relapsed ALL/LL within the confines of a Phase 1 study.

II. To assess the biologic activity of palbociclib in this patient population.

OUTLINE:

Patients receive Palbociclib PO (or via NG-tube) once daily on Days 1-21; Intrathecal cytarabine (IT ARAC) on Day 1, Doxorubicin IV push or infusion over 1-15 min on Day 4; Prednisone or prednisolone PO on days 4-31; Vincristine IV push or mini-bag per institutional policy on Days 4, 11, 18, and 25; and Pegaspargase IV over 1-2 hours on Days 5, and 18. If CNS3 leukemia is present, patients receive Intrathecal Triple Therapy (ITT) on days 4, 11,18, and 25. If CNS1 or 2 disease status, patients receive Methotrexate (IT MTX) on Days 18 and 32. Patients known to be CNS3 at study entry may receive ITT on Day 1 rather than IT ARAC. Treatment will be given for one cycle, 32 days, in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or refractory B- or T-lineage lymphoblastic leukemia and lymphoma.
* Patients with leukemia must have ≥ 5% (M2 or M3) bone marrow blasts with or without an extramedullary site of relapse. Morphologic relapse for M2 should be confirmed using flow cytometry, FISH and/or cytogenetics or molecular techniques.
* Patients with LL must have either measurable or evaluable disease.
* Patients with first or greater relapsed T-lineage ALL or LL and second or greater relapsed B-lineage ALL or LL are eligible.
* Patients with primary refractory disease with at least 2 prior induction attempts or first relapse refractory to at least one prior re-induction attempt are eligible.
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients <= 16 years of age.

  * Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately.

  1. Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. See DVL homepage for commercial and Phase 1 investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment.

     * A waiting period prior to enrollment is not required for patients receiving standard cytotoxic maintenance chemotherapy (i.e., corticosteroid, vincristine, 6MP, and/or methotrexate).
     * Intrathecal cytotoxic therapy: No waiting period is required for patients having received intrathecal cytarabine, methotrexate, and/or hydrocortisone. Intrathecal chemotherapy given at the time of diagnostic LP to evaluate for relapse prior to study enrollment is allowed.
     * At least 14 days must have elapsed after the completion of other cytotoxic therapy, with the exception of hydroxyurea, for patients not receiving standard maintenance therapy. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy.

       * NOTE: Cytoreduction with hydroxyurea in patients can be initiated and continued for up to 24 hours prior to the start of protocol therapy.
       * Note: Intrathecal chemotherapy that is given up to 72 hours prior to initiation of systemic chemotherapy per AINV18P1 counts as protocol therapy and not prior anti-cancer therapy. Intrathecal chemotherapy given > 72 hours prior does not count as protocol therapy.
  2. Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or ANC counts): >= 7 days after the last dose of agent. See DVL homepage for commercial and Phase 1 investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment.

     * NOTE: Cytoreduction with prednisone or methylprednisolone for <= 120 hours (5 days) in patients can be initiated and continued for up to 24 hours prior to the start of protocol therapy.
  3. Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody with the exception of blinatumomab, and toxicity related to prior antibody therapy must be recovered to Grade <= 1. Patients must have been off blinatumomab infusion for at least 14 days and all drug related toxicity must have resolved to Grade <= 1.
  4. Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid and toxicity related to prior immune therapy must be recovered to Grade <= 1 off corticosteroids.
  5. Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator.
  6. Interleukins, Interferons and Cytokines (other than Hematopoietic Growth Factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than Hematopoietic Growth Factors)
  7. Stem cell Infusions (with or without TBI):

     * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including DLI or boost infusion: >= 84 days after infusion and no evidence of GVHD.
     * Autologous stem cell infusion including boost infusion: >= 42 days.
  8. Cellular Therapy: >= 30 days after the completion of any type of cellular therapy (e.g. modified T cells, NK cells, dendritic cells, etc.)
  9. XRT/External Beam Irradiation including Protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial BM radiation.
  10. Patients must not have received prior exposure to palbociclib or another CDK4/6 inhibitor.
* Adequate Renal Function Defined as:

  * Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 or
  * A serum creatinine based on age/gender as follows:

    * Age: 1 to < 2 years; Male: 0.6 mg/dL; Female: 0.6 mg/dL
    * Age: 2 to < 6 years; Male: 0.8 mg/dL; Female: 0.8 mg/dL
    * Age: 6 to < 10 years; Male: 1 mg/dL; Female: 1 mg/dL
    * Age: 10 to < 13 years; Male: 1.2 mg/dL; Female: 1.2 mg/dL
    * Age: 13 to < 16 years; Male: 1.5 mg/dL; Female: 1.4 mg/dL
    * Age: >= 16 years; Male: 1.7 mg/dL; Female: 1.4 mg/dL
* Adequate Liver Function Defined as:

  * bilirubin (sum of conjugated + unconjugated) <= 1.5 x upper limit of normal (ULN) for age
  * SGPT (ALT) <= 225 U/L unless disease-related. For the purpose of this study, the ULN for SGPT is 45 U/L.
  * Serum albumin >= 2 g/dL.
* Adequate Cardiac Function Defined As:

  * Shortening fraction of >= 27% by echocardiogram, or
  * Ejection fraction of >= 50% by gated radionuclide study.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Based on the mechanism of action, palbociclib may be expected to cause fetal harm if used during pregnancy. Pregnancy tests must be obtained in girls who are post-menarche. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy. Women of reproductive potential should use effective contraception during treatment and for at least 3 weeks after the last dose of palbociclib. Males with female partners of reproductive potential should use effective contraception during treatment and for 3 months after the last dose of palbociclib. Animal data suggests that palbociclib may affect male fertility.
* Prednisone or methylprednisolone for ≤ 120 hours (5 days) may be administered for cytoreduction up to 24 hours prior to the start of protocol therapy and as treatment for allergic reactions or for physiologic replacement/stress dosing of hydrocortisone for documented adrenal insufficiency. Corticosteroids are not allowed for other indications. If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid.
* Patients who are currently receiving another investigational drug.
* Patients who are currently receiving other anti-cancer agents are not eligible [except patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy].
* Patients who are currently receiving drugs that are strong inhibitors and/or inducers of CYP3A4 or sensitive CYP3A4 substrates and CYP3A4 substrates with a narrow therapeutic range are not eligible. Strong inducers or inhibitors of CYP3A4 are prohibited from 14 days prior to enrollment to the end of the study.
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant.
* Patients must be able to swallow intact capsules or liquid. Patients that are unable to swallow oral medications may receive palbociclib through an NG tube. G tube administration is not allowed.
* Patients who have an uncontrolled infection defined as below:

  * Fever above 38.2°C within 48 hours of study enrollment with clinical signs of infection. Fever that is determined to be due to tumor burden is allowed if patients have documented negative blood cultures for at least 48 hours prior to enrollment and no concurrent signs or symptoms of active infection or hemodynamic instability.
  * A positive fungal culture within 30 days of study enrollment or active therapy for presumed invasive fungal infection.
  * Patients may be receiving IV or oral antibiotics to complete a course of therapy for a prior documented infection as long as cultures have been negative for at least 48 hours and signs or symptoms of active infection have resolved. For patients with c. difficile diarrhea, at least 72 hours of antibacterial therapy must have elapsed and stools must have normalized to baseline.
  * Active viral or protozoal infection requiring IV treatment.
* Patients known to have one of the following concomitant genetic syndromes: Down syndrome, Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachmann syndrome or any other known bone marrow failure syndrome.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Cumulative prior anthracycline exposure must not exceed 400 mg/m2 of DOXOrubicin equivalents

Ages: 12 Months to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raetz, MD, Study Chair — Children's Oncology Group
Locations (19):
- United States (19):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Raetz EA, Teachey DT, Minard C, Liu X, Norris RE, Denic KZ, Reid J, Evensen NA, Gore L, Fox E, Loh ML, Weigel BJ, Carroll WL. Palbociclib in combination with chemotherapy in pediatric and young adult patients with relapsed/refractory acute lymphoblastic leukemia and lymphoma: A Children's Oncology Group study (AINV18P1). Pediatr Blood Cancer. 2023 Nov;70(11):e30609. doi: 10.1002/pbc.30609. Epub 2023 Aug 8. PMID 37553297

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1 With 50 mg/m^2; Stratum PK With 50 mg/m^2: Patients known to be CNS3 at study entry may receive ITT on Day 1 rather than IT ARAC.
Period: Overall Study
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Started | 6 | 6
Completed | 6 | 3
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 10 [6 to 21] | 10 [6 to 13] | 10 [6 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Dose Limiting Toxicities of Palbociclib
Description: The frequency (%) of patients experiencing a cycle 1 dose limiting toxicity at least possibly attributable to Palbociclib by study part and dose level.
Time Frame: Up to 32 days
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
Participants | 1 | 0

2. Primary Outcome: Frequency of Adverse Events of Palbociclib
Description: The frequency (%) of patients experiencing adverse events at least possibly attributable to Palbociclib by study part and dose level.
Time Frame: Up to 26 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
Participants | 5 | 5

3. Primary Outcome: Area Under the Drug Concentration Curve of Palbociclib
Description: The median (min, max) of the area under the drug concentration curve for Palbociclib determined by measures at 0, 1, 2, 4, 8, and 24 hours post-dose on day 11 by study part and dose level.
Time Frame: Up to 11 days
Population: All enrolled patients
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 1278.5 [530 to 2404] | 1131.5 [486 to 1837]

4. Primary Outcome: Half-life of Palbociclib
Description: The median (min, max) of the half-life of Palbociclib determined by measures at 0, 1, 2, 4, 8, and 24 hours post-dose on day 11 by study part and dose level.
Time Frame: Up to 11 days
Population: All enrolled patients
Measure: Median (Full Range); unit: Hours
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
Hours | 23.04 [4 to 86.81] | 16.78 [4 to 39.93]

5. Primary Outcome: Maximum Serum Concentration of Palbociclib
Description: Median (min, max) of the maximum serum concentration of Palbociclib determined by measures at 0, 1, 2, 4, 8, and 24 hours post-dose on day 11 by study part and dose level
Time Frame: Up to 11 days
Population: All enrolled patients
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
ng/mL | 70.8 [31.8 to 158] | 82.15 [39.6 to 120]

6. Primary Outcome: Time to Reach Maximum Serum Concentration of Palbociclib
Description: Median (min, max) of the maximum time to reach serum concentration of Palbociclib determined by measures at 0, 1, 2, 4, 8, and 24 hours post-dose on day 11 by study part and dose level
Time Frame: Up to 11 days
Population: All enrolled patients
Measure: Median (Full Range); unit: Hours
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
Hours | 3.71 [2.08 to 8.02] | 4 [1.53 to 8.22]

7. Primary Outcome: Clearance of Palbociclib
Description: Median (min, max) of the clearance of Palbociclib determined by measures at 0, 1, 2, 4, 8, and 24 hours post-dose on day 11 by study part and dose level
Time Frame: Up to 11 days
Population: All enrolled patients
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
L/h/m^2 | 39.4 [21.1 to 93] | 42.65 [27.8 to 102]

8. Secondary Outcome: Number of Participants With at Least Partial Response to Palbociclib
Description: Frequency (%) of patients with at least partial response to Palbociclib per leukemia/lymphoma specific response criteria: Complete Response (CR), M1 marrow (<5% blasts) and absolute neutrophil count (ANC) at least 500/uL and platelet count at least 50000/uL without transfusion for 7 days; Complete response with incomplete recovery (CRi), M1 marrow (<5% blasts), ANC<500uL, platelet count <50,000uL; Partial Response (PR), Complete disappearance of circulating blasts and achievement of M2 marrow status if M3 originally, without new sites of extramedullary disease, and with ANC ≥ 500/µL. Complete response in the marrow without resolution of extramedullary sites. Overall Response (OR) = CR+CRi+PR
Time Frame: up to 26 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 6 | 6
Participants | 4 | 1

9. Secondary Outcome: Absolute Peripheral Blast Count of Palbociclib
Description: Median (min, max) of absolute peripheral blast count of palbociclib by study part and dose level
Time Frame: Up to 3 days
Population: All eligible patients
Measure: Median (Full Range); unit: peripheral blasts per microliter
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 4 | 5
peripheral blasts per microliter | 43 [7 to 97] | 54 [0 to 86]

10. Secondary Outcome: Radiographic Response of Palbociclib in Patients With LL Patients
Description: Number of LL patients with radiographic response by study part and dose level. Complete Response (CR): Disappearance of all disease; Partial Response (PR): 50% decrease in SPD (the sum of the products of the largest diameter and the perpendicular diameter for a tumor mass). Total responders = CR+PR
Time Frame: Day 32
Population: LL patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

11. Secondary Outcome: RB1 Expression of Palbociclib
Description: Median (min,max) of RB1 expression of palbociclib by study part and dose level
Time Frame: Up to 4 days
Population: Data not collected
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phospho-RB1 Expression of Palbociclib
Description: Median (min,max) of Phospho-RB1 expression of palbociclib by study part and dose level
Time Frame: Up to 4 days
Population: All eligible patients
Measure: Median (Full Range); unit: Percent of cells expressing Phospho-RB1
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 3 | 2
Percent of cells expressing Phospho-RB1 | 13 [8.4 to 19.1] | 15 [4.9 to 25.8]

13. Secondary Outcome: Cyclin D3 Expression of Palbociclib
Description: Median (min,max) of Cyclin D3 expression of palbociclib by study part and dose level
Time Frame: Up to 4 days
Population: All eligible patients
Measure: Median (Full Range); unit: mean fluorescence intensity (MFI)
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 3 | 2
mean fluorescence intensity (MFI) | 20.7 [5.14 to 26.59] | 9.6 [5.21 to 13.95]

14. Secondary Outcome: CDK4 Expression of Palbociclib
Description: Median (min,max) of CDK4 expression of palbociclib by study part and dose level
Time Frame: Up to 4 days
Population: All eligible patients
Measure: Median (Full Range); unit: mean fluorescence intensity (MFI)
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 3 | 2
mean fluorescence intensity (MFI) | 10.7 [1.5 to 10.99] | 5.8 [1.65 to 10.04]

15. Secondary Outcome: CDK6 Expression of Palbociclib
Description: Median (min,max) of CDK6 expression of palbociclib by study part and dose level
Time Frame: Up to 4 days
Population: All eligible patients
Measure: Median (Full Range); unit: mean fluorescence intensity (MFI)
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 3 | 2
mean fluorescence intensity (MFI) | 11.99 [4.26 to 15.57] | 13.96 [5.22 to 22.71]

16. Secondary Outcome: p27Kip1 Expression of Palbociclib
Description: Median (min,max) of p27Kip1 expression of palbociclib by study part and dose level
Time Frame: Up to 4 days
Population: All eligible patients. Data not collected for Stratum 1 patients.
Measure: Median (Full Range); unit: Percent of cells expressing p27kip1
Arm/Group | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 1
Percent of cells expressing p27kip1 | 11 [11 to 11]

17. Secondary Outcome: Ki67 Biological Activity of Palbociclib
Description: Median (min,max) of CD1a biological activity of palbociclib
Time Frame: Up to 32 days
Population: All eligible patients
Measure: Median (Full Range); unit: percentage of positive cells
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 3 | 2
percentage of positive cells | 0.70 [0.6 to 0.9] | 13 [3.3 to 22.8]

18. Secondary Outcome: DAPI Biological Activity of Palbociclib
Description: Median (min,max) of DAPI biological activity of palbociclib by study part and dose level
Time Frame: up to 26 months
Population: Data not collected
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 26 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Stratum 1 With 50 mg/m^2 | Stratum PK With 50 mg/m^2
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 With 50 mg/m^2 (N=6) | Stratum PK With 50 mg/m^2 (N=6)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 6
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 2 | 2
Catheter related infection (Infections and infestations) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
GGT increased (Investigations) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
INR increased (Investigations) | 0 | 1
Infections and infestations - Other, BK virus (Infections and infestations) | 1 | 0
Infections and infestations - Other, blood (Infections and infestations) | 1 | 0
Investigations - Other, Direct Bilirubin Increase (Investigations) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 5 | 5
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Multi-organ failure (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 6 | 6
Oral pain (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Platelet count decreased (Investigations) | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vitreous hemorrhage (Eye disorders) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 6 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 With 50 mg/m^2 (N=6) | Stratum PK With 50 mg/m^2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 3
Agitation (Psychiatric disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 5 | 3
Alkaline phosphatase increased (Investigations) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Anal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 4
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Blood and lymphatic system disorders - Other, Hypovolemia (Blood and lymphatic system disorders) | 0 | 1
Blood and lymphatic system disorders - Other, Hypoxemia (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac disorders - Other, (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, Bradycardia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Creatinine increased (Investigations) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ear and labyrinth disorders - Other, (Ear and labyrinth disorders) | 1 | 0
Edema limbs (General disorders) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Eye disorders - Other, (Eye disorders) | 1 | 0
Eye disorders - Other, Subconjuctival Hemorrhage (Eye disorders) | 0 | 1
Eye disorders - Other, double vision (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 1 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 1 | 4
GGT increased (Investigations) | 1 | 0
Gastrointestinal disorders - Other, Hematochezia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, Hypodense Pontine tonsillar lesion (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 1
Hypersomnia (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 3
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 6
Hypotension (Vascular disorders) | 2 | 1
INR increased (Investigations) | 0 | 1
Immune system disorders - Other, (Immune system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Investigations - Other, (Investigations) | 1 | 0
Investigations - Other, Direct Bilirubin Increased (Investigations) | 1 | 1
Investigations - Other, low total protein (Investigations) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Localized edema (General disorders) | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metabolism and nutrition disorders - Other, (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other, vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Nervous system disorders - Other, (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Papilledema (Eye disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 4
Skin and subcutaneous tissue disorders - Area below eyes w/erythema-appears like allergic shiners (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, Skin Breakdown (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Vitreous hemorrhage (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Weight gain (Investigations) | 0 | 3
Weight loss (Investigations) | 0 | 3
White blood cell decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03792256/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03792256/ICF_001.pdf